CLINICAL TRIAL: NCT07326787
Title: The Effect of a Social Cognitive Theory-Based Educational Intervention Program on Sustainable Eco-Friendly Nutrition, Nutritional Attitudes, and Self-Efficacy in Adolescents: A Randomized Controlled Trial
Brief Title: Social Cognitive Theory-Based Educational Intervention Program on Sustainable Eco-Friendly Nutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sumeyra YILMAZ, Research Assistant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: E-77082166-302.08.01-1287221
Record Dates: First submitted 2025-12-26; First posted 2026-01-08 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Sustainable Eco-Friendly Nutrition; Self Efficacy; Adolescent Nutrition
Keywords: adolescent; Sustainable Eco-Friendly Nutrition; nursing; climate change

STUDY DESIGN:
Intervention Model Description: The research will be conducted with a parallel group randomized controlled experimental design to examine the effects of a sustainable environmentally friendly nutrition educational intervention program based on social cognitive theory on sustainable environmentally friendly nutrition, nutritional attitudes, and nutritional self-efficacy in adolescents.
Who Masked: Investigator
Masking Description: To prevent selection bias in the study, adolescents will be randomly assigned to the intervention and control groups by an independent biostatistician using a simple randomization method. Adolescents will be assigned a participant number when the preliminary assessment data are transferred to the computer. The researcher will not know which group the adolescents are in until the study begins. Data will be coded and transferred to the computer without specifying the intervention and control groups. To prevent reporting bias, the study data will be evaluated by an independent biostatistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Following pretests, participants will be randomly assigned to intervention and participation groups. The intervention group will receive a total of six weeks (six sessions) of the intervention program. Each session is planned to last approximately one class hour (40 minutes). Each session will begin with presentations based on literature, followed by various activities and games to reinforce the topic and support lasting behavioral changes in students. The games were designed according to the gamification model.
  Interventions: Other: Social Cognitive Theory-Based Educational Intervention Program
- Control Group (No Intervention): The control group will not receive any intervention and will continue their education in accordance with the current curriculum. Data collection tools will be administered again one and three months after the pretest, posttest, and interventions are completed in parallel with the intervention group. The intervention may be administered after the program is completed, at the request of the school administration.

INTERVENTIONS:
Other: Social Cognitive Theory-Based Educational Intervention Program — In this study, a sustainable eco-friendly nutrition educational intervention program was developed based on social cognitive theory. The sustainable eco-friendly nutrition educational intervention program will last six weeks. Each session will consist of one session per week, covering one module. Each session is expected to last approximately 40 minutes. Each module will utilize presentations based on the content, followed by various activities and games to reinforce the topic and support lasting behavioral changes in students.
  To reinforce the knowledge and practices adolescents have learned and implemented during the program, and to strengthen the impact of the intervention, the researcher will prepare 12 SMS (Short Message Service) messages using various sources and send them individually to adolescents/parents.
  Arms: Intervention Group

SUMMARY:
This study is designed as a parallel-group randomized controlled trial to evaluate the effectiveness of a sustainable environmentally friendly nutrition educational intervention program developed based on the principles of Social Cognitive Theory. The intervention aims to improve sustainable environmentally friendly nutrition behaviors, nutritional attitudes, and nutrition self-efficacy among adolescents.

Eligible participants will be randomly assigned to either an intervention group or a control group using a computerized simple randomization procedure conducted by an independent researcher. Allocation concealment will be ensured through participant coding, and data analysis will be performed by an independent biostatistician blinded to group assignments.

The intervention group will participate in a structured six-week educational program, consisting of one session per week. Each session will last approximately 40 minutes and will focus on a specific module addressing the relationship between climate change, environmental sustainability, and nutrition. Program content is grounded in Social Cognitive Theory, emphasizing observational learning, self-regulation, outcome expectations, and self-efficacy enhancement. Educational methods will include interactive presentations, group discussions, games, and activity-based learning supported by visual and audio materials to promote engagement and long-term behavioral change.

To reinforce learning and facilitate behavior maintenance, supplementary reinforcement messages will be delivered throughout the intervention period. Communication with participants and their parents will be maintained via digital messaging platforms to support adherence and engagement.

The control group will continue their routine school curriculum without receiving any nutrition-related educational intervention during the study period.

Outcome data will be collected at four time points: baseline (pre-intervention), immediately after completion of the six-week program (post-intervention), and at one-month and three-month follow-up assessments. Data collection is expected to take approximately 25 minutes at each assessment point. The follow-up assessments are intended to evaluate the sustainability of behavior change over time.

The intervention will be implemented during the fall semester of the 2025-2026 academic year following the completion of ethical approval and institutional permissions.

DETAILED DESCRIPTION:
This study is designed as a parallel-group randomized controlled trial to evaluate the effectiveness of a sustainable environmentally friendly nutrition educational intervention program developed based on the principles of Social Cognitive Theory. The intervention aims to improve sustainable environmentally friendly nutrition behaviors, nutritional attitudes, and nutrition self-efficacy among adolescents.

Eligible participants will be randomly assigned to either an intervention group or a control group using a computerized simple randomization procedure conducted by an independent researcher. Allocation concealment will be ensured through participant coding, and data analysis will be performed by an independent biostatistician blinded to group assignments.

The intervention group will participate in a structured six-week educational program, consisting of one session per week. Each session will last approximately 40 minutes and will focus on a specific module addressing the relationship between climate change, environmental sustainability, and nutrition. Program content is grounded in Social Cognitive Theory, emphasizing observational learning, self-regulation, outcome expectations, and self-efficacy enhancement. Educational methods will include interactive presentations, group discussions, games, and activity-based learning supported by visual and audio materials to promote engagement and long-term behavioral change.

To reinforce learning and facilitate behavior maintenance, supplementary reinforcement messages will be delivered throughout the intervention period. Communication with participants and their parents will be maintained via digital messaging platforms to support adherence and engagement.

The control group will continue their routine school curriculum without receiving any nutrition-related educational intervention during the study period.

Outcome data will be collected at four time points: baseline (pre-intervention), immediately after completion of the six-week program (post-intervention), and at one-month and three-month follow-up assessments. Data collection is expected to take approximately 25 minutes at each assessment point. The follow-up assessments are intended to evaluate the sustainability of behavior change over time.

The intervention will be implemented during the fall semester of the 2025-2026 academic year following the completion of ethical approval and institutional permissions.

ELIGIBILITY:
Inclusion Criteria:

* Being a 6th or 7th grade student
* Volunteering to participate in the study
* Family approval for participation in the study

Exclusion Criteria:

* Following a specific nutrition program
* Having communication difficulties (hearing, seeing, or understanding)
* Having plans to travel/move out of town during the work period
* Having special needs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-09-22 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Child Nutrition Self-Efficacy Scale | Pre-intervention (week 1), post-intervention (week 6), follow-up time (at the end of month 1 and 3)
  It was measured with the "Child Nutrition Self-Efficacy Scale", which is used to evaluate children's self-efficacy regarding nutrition. The scale consists of 15 items rated on a 3-point Likert scale. Total scores range from -15 to +15, with higher scores indicating greater nutrition self-efficacy and healthier food choices.
"Sustainable Eco-Friendly Nutrition Scale | Pre-intervention (week 1), post-intervention (week 6), follow-up time (at the end of month 1 and 3)
  The "Sustainable Eco-Friendly Nutrition Scale," developed by the researcher, was used to assess participants' sustainable eco-friendly nutritional behaviors. Higher scores on the scale indicate increased sustainable eco-friendly nutritional behavior The scale consists of 19 items rated on a 5-point Likert scale. Total scores range from 19 to 95, with higher scores indicating higher levels of sustainable environmentally friendly nutrition behavior.
Nutrition Attitude Subscale | Pre-intervention (week 1), post-intervention (week 6), follow-up time (at the end of month 1 and 3)
  It was measured with the "Nutrition Attitude Subscale" used to determine the participants' attitudes towards healthy nutrition. The nutrition subscale consists of 4 items rated on a 4-point Likert scale. Total scores range from 4 to 16, with higher scores indicating more positive nutrition attitudes.

CONTACTS AND LOCATIONS:
Overall Officials: Sümeyra Yılmaz, Principal Investigator — Gazi University
Locations (1):
- Secondary School, Ankara, Turkey (Türkiye)